CLINICAL TRIAL: NCT02836327
Title: Multimodel MRI to Explore the Pathophysiology of Multiple Sclerosis and Neuromyelitis Optica Spectrum Disorders
Brief Title: Multimodel Magnetic Resonance Imaging (MRI)of Multiple Sclerosis and Neuromyelitis Optica Spectrum Disorders
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Xin Lou, Deputy Chief, Chinese PLA General Hospital
Other Study IDs: MS and NMOSD-ChinaPLAGH
Record Dates: First submitted 2016-07-14; First posted 2016-07-19 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Multiple Sclerosis; Neuromyelitis Optica Spectrum Disorders
Keywords: MRI; Multiple Sclerosis; Neuromyelitis Optica Spectrum Disorders; Multimodel
MeSH Terms: conditions — Multiple Sclerosis; Neuromyelitis Optica | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Multiple sclerosis: Multiple sclerosis patients confirmed by neurologist according to the 2010 revised Mcdonald criteria without other nervous system diseases.All patients performed magnetic resonance imaging.
  Interventions: Other: Magnetic Resonance Imaging
- Neuromyelitis optica spectrum disorders: Neuromyelitis optica spectrum disorders confirmed by neurologist according to the 2015 revised diagnostic criteria without other nervous system diseases.All patients performed magnetic resonance imaging.
  Interventions: Other: Magnetic Resonance Imaging
- Health control: Health control is defined as no other nervous system diseases such as ischemic stroke, alzheimer disease and so on. The baseline data(age,education background etc.) is similar to multiple sclerosis and neuromyelitis optica spectrum disorders patients.All participants performed magnetic resonance imaging.
  Interventions: Other: Magnetic Resonance Imaging

INTERVENTIONS:
Other: Magnetic Resonance Imaging — Magnetic Resonance Imaging

SUMMARY:
To investigate multimodel MRI exploring the pathophysiology of multiple sclerosis and neuromyelitis optica spectrum disorders.

The investigators use multimodel MRI to evaluate the extent of blood-brain barrier and white matter fiber tracts destruction , iron deposition and cerebral blood flow of associated regions in multiple sclerosis and neuromyelitis optica spectrum disorders using contrast-enhanced magnetic resonance imaging , quantitative susceptibility mapping, diffusion tension imaging, and arterial spin labeling with post labeling delay of 2.0 seconds. Transfer constant volume , magnetic susceptibility, cerebral blood flow and fractional anisotropy(FA) value were measured in lesion and normal appearing white matter.

DETAILED DESCRIPTION:
Patients:

Patients with multiple sclerosis and neuromyelitis optica spectrum disorders were included. clinical characteristics such as disease duration, expanded disability status scale(EDSS) score, age, associated laboratory examination(autoantibodies directed to aquaporin-4 and oligoclonal bands in serum as well as cerebrospinal fluid)were recorded.

Imaging scan were conducted at admission, six months and one year after admission

Imaging protocols:

MRI scan protocols: T2 weighted image, T1 weighted image, Diffusion weighted image(DWI), fluid-attenuated inversion recovery(FLAIR), dynamic contrast-enhanced magnetic resonance imaging(DCE-MRI) , diffusion tension imaging(DTI) ,quantitative susceptibility mapping(QSM) , arterial spin labeling(ASL) with post labeling delay(PLD) of seconds, sagittal CUBE Fluid Attenuation Inversion Recovery (FLAIR) images, sagittal 3-dimensional Fast Spoiled Gradient Echo(3D-FSPGR).

Contrast agent:

Omniscan 0.1mmol/kg, Inject rate：2ml/s

Imaging evaluation:

Transfer constant volume value measured by DCE-MRI indicates the extent of blood-brain barrier destruction.

Magnetic susceptibility manifests iron deposition in lesions and normal appearing white matter.

Diffusion tension imaging demonstrates the extent of white matter fiber tracts destruction.

Arterial spin labeling(ASL) with post labeling delay(PLD)of seconds shows cerebral blood flow in associated regions.

ELIGIBILITY:
Inclusion Criteria:

1. a diagnosis of neuromyelitis optica spectrum disorders(according to the 2015 revised diagnostic criteria) or relapsing remitting multiple sclerosis(according to the 2010 revised Mcdonald criteria)
2. age between 18 years old and 60 years old(concluding 18 years old and 60 years old)

Exclusion Criteria:

1. common exclusion for MRI such as patients with claustrophobia
2. patients with poor imaging quality（Poor imaging quality mainly defined as the image cannot be applied to future analysis on account of severe motion artifacts appeared in conventional MRI and mistakes in the MRI process by accident factors which cannot to be applied to future analysis）
3. patients with taking amount of antidepressant recently and with alcoholism and other nervous system diseases

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: patients with multiple sclerosis (according to the 2010 revised Mcdonald criteria) and neuromyelitis optica spectrum disorders (according to the 2015 revised diagnostic criteria)
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2014-09; Primary Completion 2019-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Recurrence | three months to one year
  The patients will be monitored whether they recured multiple sclerosis and neuromyelitis optica spectrum disorders confirmed by neurologist and conventional MRI.
  Clinical suspicious signs of recurrence : visual loss,urination and defecation function disturbance and so on.
  Conventional MRI: there are new lesions or the lesions show high signal on diffusion weighted images or enhancement on post contrast enhanced images.

CONTACTS AND LOCATIONS:
Overall Officials: Xin Lou, M.D.,Ph.D., Study Chair — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided